CLINICAL TRIAL: NCT06803303
Title: Added Value of Sonoelastography in Assessment of Traumatic and Non Traumatic Supraspinatus Tendinopathy and Tear Compared with Magnetic Resonance Imaging
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Hassan Sayed, doctor, Assiut University
Other Study IDs: supraspinatus sonoelastography
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Supraspinatus Injury
Keywords: Supraspinatus sonoelastography
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: sonoelastography — Sonoelastography examination[10,11] will be performed using (GE logiqs8,) device system with a high-frequency (a 5-12 MHz linearMHz) linear probe. The procedure will be carried out by a radiologist , who is blinded to the MRI results.
  Magnetic resonance imaging (MRI) [12] will be performed on the patients in our radiology department using a Philips Achieva 1.5 Tesla superconducting magnet (The Netherlands), shoulder joint MRI protocol included several imaging sequences, included coronal oblique T1 and T2 weighted fast spin-echo, coronal oblique proton density fat suppressed, oblique sagittal T2-weighted spin-echo and axial T1-weighted spin-echo Image evaluation will be conducted by experienced musculoskeletal radiologist, Then we correlate results of sonoelastography to that of MRI .

SUMMARY:
Primary Aims:

To assess the value of sonoelastography in the evaluation of supraspinatus tendon abnormalities.

Secondary Aims:

1. To assess the association between SWE and grades of tendon abnormalities on MRI (the standard imaging in the evaluation of rotator cuff abnormalities).
2. To help in reaching shear wave elastography cutoff value to determine tendinopathy and tear.

DETAILED DESCRIPTION:
Shoulder pain is a common condition that can be caused by a variety of factors, including injury, overuse, poor posture, and age-related degeneration. The shoulder is a highly mobile joint, which makes it prone to certain injuries and conditions. The pain can arise from structures in or around the shoulder joint, including the muscles, tendons, ligaments, and the bones of the shoulder itself.

Rotator cuff abnormalities one of the important causes that can cause chronic shoulder pain , discomfort and lead to a lack of stability of the shoulder joint[1].The supraspinatus tendon is one of rotator cuff muscle that commonly affected as it anatomically traverses between two bones (the acromion process and humeral head),its pathology including tendinopathy and tearing whether its partial or complete.

Clinical examination and imaging modalities as ultrasound and MRI are needed for proper diagnosis of supraspinatus pathology .

Ultrasonography used as primary modality compared to MRI which considered gold standard of non invasive investigations as ultrasound is an cheap, available, noninvasive, repeatable and reliable modality for rotator cuff assessment with accuracy reaching 100% in the diagnosis of full-thickness tears and 91% for partial-thickness tears, on ultrasound, tendinopathy appears as thickening of the tendon showing a heterogeneous hypoechoic pattern. Tendon tear appears as a hypoechoic defect within the tendon, not involving the tendon's full thickness in PTT and involving the full tendon thickness in FTT , however, diagnosis of tendinopathy may be challenging with the conventional US as the echogenicity of the affected tendon may appear similar to that of the healthy one, especially in early stages of tendinopathy.

Sonoelastography (SE) is a new US imaging technique that allows non invasive estimation of tissue stiffness and elasticity. It is based on the fact that tissue compression produces displacement within the tissue, which is less in hard than in soft tissue [8], In addition possibility of using share wave elastography which allow to assess tissue stiffness by measuring the propagation speed of shear waves in the body. It is primarily used to evaluate the stiffness of tissues such as muscles, liver, and tendons, aiding in differentiation between the diseased and normal tissue, as tendon softening in cases of tendinopathy, resulting in a reduction in the velocity of propagation of shear waves compared to the healthy tendons that are stiff, so elastography may be helpful in the early detection of tendinopathy before alteration in tendon echogenicity or thickness appear on the conventional US. And provides qualitative as well as quantitative assessment of tendon quality through alteration in the tissue composition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with shoulder pain either due to traumatic or non traumatic causes
* Age > 18 year

Exclusion Criteria:

* History of operative intervention for rotator cuff tendons,
* Signs of calcific tendinopathy on MRI or ultrasound (as calcification causes artifact on obtaining SWE results and the measured velocities were exceeding the velocity scale on our device),
* Patients with general contraindications to MRI as patients with pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with shoulder pain either due to traumatic or non traumatic causes referred to our radiology department for assessment of rotator cuff muscles.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To assess the value of sonoelastography in the evaluation of supraspinatus tendon abnormalities | 2 year
  Assess the value of sonoelastography in evaluation of supraspinatus tendinopathy and tear in comparison with Magnetic Resonance Imaging

SECONDARY OUTCOMES:
1. To assess the association between share wave elastography and grades of tendon abnormalities on MRI (the standard imaging in the evaluation of rotator cuff abnormalities). | 2 year
2. To help in reaching shear wave elastography cutoff value to determine tendinopathy and tear | 2 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sein ML, Walton J, Linklater J, Harris C, Dugal T, Appleyard R, Kirkbride B, Kuah D, Murrell GA. Reliability of MRI assessment of supraspinatus tendinopathy. Br J Sports Med. 2007 Aug;41(8):e9. doi: 10.1136/bjsm.2006.034421. Epub 2007 Feb 8. PMID 17289860
- [Background] Jacobson JA. Shoulder US: anatomy, technique, and scanning pitfalls. Radiology. 2011 Jul;260(1):6-16. doi: 10.1148/radiol.11101082. PMID 21697306
- [Background] Amr A. Elfattah Hassan Gadalla, Gehad Ramadan Hassanein, Hatem Mohammed Saeed El Azizy, Walid Reda Mohammed & Neiven Ezzat Mohammed Elliethy ,Egyptian Journal of Radiology and Nuclear Medicine volume 54, Article number: 37 (2023) Cite this articl
- [Background] Reem A. Frere a, Ibrahim Libda a, Fathy Tantawy a, Hossam M. Sakr b, Ali T. El-Alfy, Sonoelastography, conventional ultrasound and magnetic resonance imaging in detection of rotator cuff lesions in patients with chronic shoulder pain, The Egyptian Rheumatologist,Volume 43, Issue 1, January 2021, Pages 17-21
- [Background] Winn N, Lalam R, Cassar-Pullicino V. Sonoelastography in the musculoskeletal system: Current role and future directions. World J Radiol. 2016 Nov 28;8(11):868-879. doi: 10.4329/wjr.v8.i11.868. PMID 27928468
- [Background] Manzoor I, Bacha R, Gilani SA. Diagnostic accuracy of sonoelastography in different diseases. J Ultrason. 2018 Mar;18(72):29-36. doi: 10.15557/JoU.2018.0005. Epub 2018 Mar 30. PMID 29844938
- [Background] Seo JB, Yoo JS, Ryu JW. Sonoelastography findings of supraspinatus tendon in rotator cuff tendinopathy without tear: comparison with magnetic resonance images and conventional ultrasonography. J Ultrasound. 2014 Dec 7;18(2):143-9. doi: 10.1007/s40477-014-0148-8. eCollection 2015 Jun. PMID 26191102
- [Background] Vlychou M, Dailiana Z, Fotiadou A, Papanagiotou M, Fezoulidis IV, Malizos K. Symptomatic partial rotator cuff tears: diagnostic performance of ultrasound and magnetic resonance imaging with surgical correlation. Acta Radiol. 2009 Jan;50(1):101-5. doi: 10.1080/02841850802600764. PMID 19052931
- [Background] Shin KM. Partial-thickness rotator cuff tears. Korean J Pain. 2011 Jun;24(2):69-73. doi: 10.3344/kjp.2011.24.2.69. Epub 2011 Jun 3. PMID 21716613
- [Background] Bendale S, Vedpathak S (2019) Sonographic Evaluation of rotator cuff pathologies causing restricted movements of shoulder. Int J Contemp Med Surg Radiol 4(3):C276-C280
- [Background] Tawfik AM, El-Morsy A, Badran MA. Rotator cuff disorders: How to write a surgically relevant magnetic resonance imaging report? World J Radiol. 2014 Jun 28;6(6):274-83. doi: 10.4329/wjr.v6.i6.274. PMID 24976930